CLINICAL TRIAL: NCT01458769
Title: Open-labeled, Randomized, Crossover, Single-dose Study in Healthy Male Subjects to Evaluate the Pharmacokinetics, Safety & Tolerability of Stable Isotopologs of Atazanavir (ATV), Administered as Single Agents or as Combinations of Two Isotopologs, With a Pharmacokinetic Comparison to Reyataz®.
Brief Title: Pharmacokinetics, Safety & Tolerability of Isotopologs of Atazanavir (ATV), With Pharmacokinetic Comparison to Reyataz
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Concert Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CP405.1003
Record Dates: First submitted 2011-06-22; First posted 2011-10-25 (Estimated); Last update posted 2013-05-24 (Estimated); Status verified 2013-05

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Atazanavir Sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- Part A1 (Active Comparator): Part A1 will evaluate two single ascending doses of the single agent C-10276 (an ATV isotopolog), and a dose of Reyataz.
  C-10276 200 mg -> C-10276 400 mg -> Reyataz 400 mg
  C-10276 200 mg -> Reyataz 400 mg -> C-10276 400 mg
  Interventions: Drug: C-10276
- Part A2 (Active Comparator): Part A2 will evaluate the single agent C-10276, co-administration of CTP-518 and C-10276, and a dose of Reyataz.
  C-10276 300 mg -> Co-dose Ratio 1 CTP-518 (100 mg) with C-10276 (300 mg)-> C-10276 400 mg
  C-10276 300 mg -> C-10276 400 mg -> Co-dose Ratio 1 CTP-518 (100 mg) with C-10276 (300 mg)
  Interventions: Drug: C-10276
- Part B Group 1 (Active Comparator): Group B1 will evaluate single doses of an ATV isotopolog, C-10297.
  C-10297 200 mg
  Interventions: Drug: C-10297
- Part B Group 2 (Active Comparator): Group B2 will evaluate single doses of an ATV isotopolog, C-10299.
  C-10299 200 mg
  Interventions: Drug: C-10299
- Part B Group 3 (Active Comparator): Group B3 will evaluate two single ascending doses of isotopologs C-10297 and 400 mg dose of Reyataz in a 3-way crossover design.
  C-10297 400 mg -> Reyataz 400 mg -> C-10297 600 mg
  Interventions: Drug: C-10297; Drug: Reyataz®
- Part B Group 4 (Active Comparator): Group B4 will evaluate two single ascending doses of isotopolog C-10299 and a 400 mg dose of Reyataz in a 3-way crossover design.
  C-10299 400 mg -> Reyataz 400 mg -> C-10299 600 mg
  Interventions: Drug: C-10299; Drug: Reyataz®
- Part B Group 5 (Active Comparator): Group B5 will evaluate a single dose of C-10276 and a 400 and 600 mg dose of Reyataz in a 3-way crossover design.
  C-10276 600 mg -> Reyataz 400 mg -> Reyataz 600 mg
  Interventions: Drug: C-10276; Drug: Reyataz®

INTERVENTIONS:
Drug: C-10276 — C-10276 200 mg, C-10276 400 mg, Reyataz 400 mg oral, single dose
  Arms: Part A1
Drug: C-10276 — C-10276 300 mg, CTP-518 100 mg with C-10276 300 mg, C-10276 400 mg oral, single dose
  Arms: Part A2
Drug: C-10297 — C-10297 200 mg, oral, single dose
  Arms: Part B Group 1
Drug: C-10299 — C-10299 200 mg, oral, single dose
  Arms: Part B Group 2
Drug: C-10297 — C-10297 400 mg, Reyataz 400 mg, C-10297 600 mg, oral, single dose
  Arms: Part B Group 3
Drug: C-10299 — C-10299 400 mg, Reyataz 400 mg, C-10299 600 mg, oral, single dose
  Arms: Part B Group 4
Drug: C-10276 — C-10276 600 mg, Reyataz 400 mg, Reyataz 600 mg, oral, single dose
  Arms: Part B Group 5
Drug: Reyataz® — Reyataz 400 mg, oral, single dose Reyataz 600 mg, oral, single dose
  Arms: Part B Group 3; Part B Group 4; Part B Group 5

SUMMARY:
The purpose of this study is to assess the safety, tolerability and pharmacokinetics of isotopologs of Atazanavir both as single agents and as combinations.

DETAILED DESCRIPTION:
There are two parts to this study. Part A is a three-period, crossover design. Eligible subjects will be randomized to 1 of 4 sequences, in groups of 4 subjects each. All study drug doses, including the comparator, Reyataz, will be administered as single, open-labeled doses to subjects after a light meal. There will be a 7-day washout between individual subjects doses; that is, dosing will occur on the same day each week.

Part B evaluations are based on the results of Part A. Part B will further consist of two subparts. In the first subpart, low single doses of 2 new isotopologs will be dosed to two groups of 4 subjects each, B1 and B2, respectively. Following assessment of safety and pharmacokinetics in the first subpart, the second subpart, which consists of three groups of 8 subjects (B3, B4, B5) each will be dosed. Subjects enrolled in B3, B4, and B5 will participate in a 3-way partial crossover study design.

The objectives will be to compare the PK properties, in healthy male subjects after a light meal, of single oral doses of single agent ATV isotopologs or as combinations of two ATV isotopologs with the PK properties in the same subjects, after a light meal, of a single dose of either 400 mg or 600 mg Reyataz. The safety and tolerability will also be evaluated.

Blood samples for pharmacokinetic analysis will be collected. Actual dosing and sampling times will be used for analysis.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, as determined by the responsible physician, based on a medical evaluation including history, physical examination, vital signs, electrocardiograms (ECGs) and laboratory tests assessed at the screening visit and prior to the first dose of study drug. A subject with a non-clinically significant abnormality or laboratory parameters outside the reference range may be included only if the investigator considers that the finding will not compromise the subject's safety and will not interfere with the study procedures or data interpretation.
* Healthy adult males between 18 and 50 years of age, inclusive
* Body weight ≥ 50 kg and BMI within the range of 18 to 32 kg/m2, inclusive, at screening
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form and the protocol
* Willing and able to be confined at the clinical research center for the study days
* Negative tests for selected drugs of abuse, cotinine, and alcohol at screening and Day -1
* Dietary habits that fall within the range of normal, as determined by the investigator. Examples of unusual diets are liquid diets, protein-only diets, high fat-diets, or low-carbohydrate diets.
* Willingness of male subjects to abstain from sexual intercourse with pregnant or lactating women; and if engaging in sexual intercourse with a female partner who could become pregnant, a willingness of male subjects to use a condom and spermicide, in addition to having the female partner use another form of contraception such as an intrauterine device, diaphragm with spermicide, oral contraceptives, injectable progesterone, subdermal implants, or a tubal ligation. This criterion must be followed from the time of first study drug administration until 30 days after the final administration of study drug.

Exclusion Criteria:

* History of clinically significant central nervous system (eg, seizures), cardiac, pulmonary, metabolic, renal, hepatic, or gastrointestinal (GI) conditions; or history of such conditions that, in the opinion of the investigator, may place the subject at an unacceptable risk as a participant in this trial, may interfere with the interpretation of safety and/or tolerability data obtained in the trial, or may interfere with the absorption, distribution, metabolism, or excretion of the study drugs
* PR interval ≥ 220 msec or QRS duration ≥ 120 msec or QT interval > 450 msec obtained at screening visit or prior to the first dose of study drug
* Aspartate transaminase (AST), alanine transaminase (ALT), gamma-glutamyl transferase (GGT), serum creatinine, or bilirubin > upper limit of normal (ULN) at screening or prior to the first dose of study drug. These laboratory tests may be repeated once, if they are abnormal on first screening, and if there is a medical reason to believe the results may be inaccurate. If the repeat test is within the reference range, the subject may be included only if the investigator considers that the previous finding will not compromise the subject's safety and will not interfere with the interpretation of safety data.
* Positive blood screen for human immunodeficiency virus (HIV antibody), hepatitis B virus surface antigen, or hepatitis C virus antibody at screening
* Urinalysis positive for protein or glucose (greater than trace findings of protein or glucose) at screening or prior to the first dose of study drug
* History of drug abuse within 6 months of screening
* History of any tobacco product use within 3 months prior to the study, to be verified by a urine cotinine screen of < 200 ng/mL at screening and prior to the first dose of study drug
* Participation in a clinical trial and receipt of an investigational medication or a new chemical entity within 30 days, 5 half-lives, or twice the duration of the biological effect of any medication (whichever is longer) prior to the first dose of current study drug
* Use of prescription or non-prescription medications, including herbal and dietary supplements within 7 days or 5 half-lives (whichever is longer) prior to the first dose of study drug, or use of St. John's Wort within 14 days prior to the first dose of study drug. (The subject may take paracetamol (≤ 2 grams/day) or ibuprofen (≤ 1600 mg/day) for up to 48 hours prior to the first dose of study drug. The investigator and study team may review medication use on a case-by-case basis to determine if its use would compromise subject safety or interfere with study procedures or data interpretation.)
* Consumption of grapefruit, grapefruit juice, star fruit, oranges, orange juice, Seville oranges, or red wine within 7 days prior to administration of study drug
* Consumption of any caffeine and/or xanthine products (ie, coffee, tea, chocolate and caffeine containing sodas, colas, etc) within 48 hours prior to each dose of study drug and while confined at the clinical site
* Donation of blood or blood products or blood collection in excess of 470 mL within 8 weeks prior to dosing
* History of sensitivity to any of the study drugs or components thereof, or a history of medication allergy or other allergy that, in the opinion of the investigator, contraindicates study participation
* Unwillingness to comply with protocol-specified lifestyle and/or dietary restrictions
* Major surgery within 4 weeks of screening
* Uncontrolled intercurrent illness (ie, active infection)
* Any other medical or psychiatric illness that could, in the investigator's opinion, compromise the subject's safety or interfere with the completion of this protocol

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2010-12; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Profile of Pharmacokinetics | predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16, 24, 30, 36,48 hours
  AUC, Cmax, C24

SECONDARY OUTCOMES:
Safety | 3 days
  Number of adverse events, change in laboratory parameters, changes from baseline in blood pressure and ECGs

CONTACTS AND LOCATIONS:
Overall Officials: Sepehr Shakib, MD, Principal Investigator — Adelaide, SA 5000 Australia